CLINICAL TRIAL: NCT03501654
Title: Prospective Clinical Trial of Unilateral or Bilateral Implantation of the Enlarged Depth-of-focus Intraocular Lens in Cataract Patients With Presbyopia
Brief Title: Prospective Clinical Trial of Unilateral or Bilateral Implantation of TecnisSymfony IOL in Cataract Patients With Presbyopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Mee Kum Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TecnisSymfony Trial
Record Dates: First submitted 2018-03-14; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Cataract; Presbyopia
Keywords: Lenses, Intraocular
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TecnisSymfony intraocular lens insertion group (Experimental)
  Interventions: Device: TecnisSymfony®

INTERVENTIONS:
Device: TecnisSymfony® — Patients received implantation of unilateral or bilateral TecnisSymfony® IOL after phacoemulsification by a single surgeon (MK Kim).

SUMMARY:
This is to evaluate the satisfaction of patient and physician about short-distance, medium-distance, long-distance postoperative vision and eyeglass dependence, glare, and visual acuity after insertion of the TECNIS® Symfony or TECNIS® Symfony Toric intraocular lens.

DETAILED DESCRIPTION:
The patients underwent uneventful phacoemulsification and implantation of TecnisSymfony®. Mean absolute error (MAE) at 1 month was compared in SRK/T, Holladay2, Haigis, Hoffer Q, Barrett Universal II, and Hill-RBF formula. At postoperative 1, 4, and 12 weeks, logMAR visual acuity (logMARVA) at the distance (5m), intermediate (66cm), and near (40cm), and spherical equivalent (SE) in manifested refraction (MR) and automated refraction (AR) were measured. Wavefront aberration, contrast sensitivity test, and glare test were done at 12 weeks. The questionnaire was used to investigate glare, glasses dependency, and patient satisfaction at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral or bilateral cataract
* Sixteen years and older
* Regular corneal topography and corneal astigmatism
* Corneal astigmatism 0.75 Diopter and less for TECNIS® Symfony IOL, and between 1.0 and 3.62 Diopter for TECNIS® Symfony toric IOL

Exclusion Criteria:

* Pregnant or nursing women
* In the presence of other ocular diseases that may affect the stability of the lens capsule (pseudoexfoliation syndrome, glaucoma, traumatic cataract, Malfan syndrome, etc.)
* White cataract
* Patients who need intraocular lens outside of range
* In the presence of other ocular diseases that is expected to have a poor final visual acuity of less than 20/30 after surgery (amblyopia, strabismus, keratoconus, etc.)
* Pupil abnormality (non-reactive pupil, tonic pupils, abnormally shaped pupils, etc.)
* Patients using systemic or ocular medication that affect visual acuity.
* Patients who had previously undergone refractive surgery.
* Patients participating in other clinical trials during the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change of visual acuity at near, intermediate and far | preoperative(last outpatient follow-up before the surgery), 1 month after surgery, 3 months after surgery.
  LogMAR visual acuity (logMARVA) at the distance (5m), intermediate (66cm), and near (40cm) were measured at preoperative (last outpatient follow-up before the surgery), postoperative 1, 4, and 12 weeks.

SECONDARY OUTCOMES:
Photic phenomena evaluation by questionnaire. | One month and three months after the surgery.
  Patients were asked if they had subjective glare or halo (scale: mild, moderate, severe).
Spectacle dependence evaluation by questionnaire | One month and three months after the surgery.
  Patients were asked for 0, 25, 50, 75, and 100% of the need to wear glasses at distance, mid-range, and near distance.

CONTACTS AND LOCATIONS:
Overall Officials: Mee Kum Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No